CLINICAL TRIAL: NCT06733532
Title: Comparison of the Beverage Hydration Index of Different Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2024-372
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hydration

STUDY DESIGN:
Intervention Model Description: semi-blinded
Who Masked: Participant
Masking Description: treatments labeled A-C. Subjects will be provided the beverage in plastic cups without product labels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Propel, Essentia, Smart (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will consume the assigned treatment (one treatment per visit in order state in arm title) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Berry Propel Fitness Water; Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate; Dietary Supplement: Smart Water
- Propel, Smart, Essentia (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will consume the assigned treatment (one treatment per visit in order state in arm title) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Berry Propel Fitness Water; Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate; Dietary Supplement: Smart Water
- Essentia, Smart, Propel (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will consume the assigned treatment (one treatment per visit in order state in arm title) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Berry Propel Fitness Water; Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate; Dietary Supplement: Smart Water
- Essentia, Propel, Smart (Active Comparator): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will consume the assigned treatment (one treatment per visit in order state in arm title) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Berry Propel Fitness Water; Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate; Dietary Supplement: Smart Water
- Smart, Essentia, Propel (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will consume the assigned treatment (one treatment per visit in order state in arm title) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Berry Propel Fitness Water; Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate; Dietary Supplement: Smart Water
- Smart, Propel, Essentia (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will consume the assigned treatment (one treatment per visit in order state in arm title) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Berry Propel Fitness Water; Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate; Dietary Supplement: Smart Water

INTERVENTIONS:
Dietary Supplement: Berry Propel Fitness Water — Subject will consume 1 Liter of commercially available Berry Propel Fitness Water at a rate of 250 milliliters per 7.5 minutes
Dietary Supplement: Essentia Hydroboost Raspberry Pomegranate — Subject will consume 1 Liter of commercially available Essentia Hydroboost Raspberry Pomegranate at a rate of 250 milliliters per 7.5 minutes
Dietary Supplement: Smart Water — Subject will consume 1 Liter of commercially available Smart Water at a rate of 250 milliliters per 7.5 minutes.

SUMMARY:
The present study will assess the effects of two different hydration solutions compared to water on hydration measures. It will follow the same approach as used by Maughan and colleagues (2016) to measure the fluid balance (the difference between the amount of water consumed and passed as urine) and beverage hydration index (the relative amount of urine passed after consumption of a drink compared to water) including time in positive fluid balance. Additionally, hydration status will be assessed with mood and digestive health questionnaires and blood pressure urine electrolyte concentrations, specific gravity, and osmolality determinations. The two oral rehydration solutions (Berry Propel Fitness Water and Essentia Hydroboost Raspberry Pomegranate) will be compared to the control (Smart Water). The purpose is to assess whether the changes in beverage composition improve the BHI above water alone for both treatments, with an hypothesized greater improvement in BHI observed with the Essentia Hydroboost Raspberry Pomegranate, due to the addition of carbohydrate.

DETAILED DESCRIPTION:
The present study will assess the effects of two different hydration solutions compared to water on hydration measures. It will follow the same approach as used by Maughan and colleagues (2016) to measure the fluid balance (the difference between the amount of water consumed and passed as urine) and beverage hydration index (the relative amount of urine passed after consumption of a drink compared to water) including time in positive fluid balance. Additionally, hydration status will be assessed with mood and digestive health questionnaires and blood pressure urine electrolyte concentrations, specific gravity, and osmolality determinations. The two oral rehydration solutions (Berry Propel Fitness Water and Essentia Hydroboost Raspberry Pomegranate) will be compared to the control (Smart Water). The purpose is to assess whether the changes in beverage composition improve the BHI above water alone for both treatments, with an hypothesized greater improvement in BHI observed with the Essentia Hydroboost Raspberry Pomegranate, due to the addition of carbohydrate.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) <35 kg/m2 (not morbidly obese)
* Cannot have a sensitivity or be allergic to any components of the study product they will be excluded.
* non-tobacco user
* cannot be following a specialized dietary pattern that may alter findings (e.g., low carbohydrate/ketogenic diet, carnivore diet, intermittent fasting etc.)
* willing to replicate the same dietary intake/activity (exercise) level for each day before a lab visit excluding screening
* Will consume a minimum of 2 liters (women) or 2.5 liters (men) of water per day, on each day prior to experimental lab visits (excluding screening)
* Will arrive to lab for visits euhydrated (USG 1.005-1.020)
* Will not consume alcohol-containing beverages within 24 hours of testing
* Will not consume caffeine-containing beverages within 12 hours of testing
* can fast (consume water/treatments only) for 15 hours (10 hours prior to lab visits not including screening)
* avoid strenuous activity for 24 hours prior to study visits excluding screening
* Will not have a history or presence of a clinically relevant (that required or requires treatment) cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder (reviewed by Nurse practitioner)
* Will not have other conditions that is likely to alter fluid balance or be negatively affected by changing electrolyte levels/hydration status (as determined by Nurse practitioner)
* Is not consuming any medication which may alter fluid retention/electrolyte levels such as sodium-glucose co-transporter 2 (SGLT2) inhibitor (for type 2 diabetes), laxatives, diuretics, Apremilast, chemotherapy, or lithium. (Medications will be reviewed by Nurse practitioner)
* Will not consume nutritional supplements, performance enhancing drugs, and/or non-steroidal anti-inflammatory drugs within 7 days of study visits excluding screening.
* cannot be enrolled in another clinical study within 30 days of the first study visit
* without active infection or illness of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Beverage Hydration Index | 0 minutes after beverage consumption
  Beverage Hydration Index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment
Beverage Hydration Index | 60 minutes after beverage consumption
  Beverage Hydration Index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment
Beverage Hydration Index | 120 minutes after beverage consumption
  Beverage Hydration Index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment
Beverage Hydration Index | 180 minutes after beverage consumption
  Beverage Hydration Index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment
Beverage Hydration Index | 240 minutes after beverage consumption
  Beverage Hydration Index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment

SECONDARY OUTCOMES:
Net Fluid Balance | 0 minutes after beverage consumption
  Net fluid balance will be calculated subtracting the total urine collected from the total liquid consumed
Net Fluid Balance | 60 minutes after beverage consumption
  Net fluid balance will be calculated subtracting the total urine collected from the total liquid consumed
Net Fluid Balance | 120 minutes after beverage consumption
  Net fluid balance will be calculated subtracting the total urine collected from the total liquid consumed
Net Fluid Balance | 180 minutes after beverage consumption
  Net fluid balance will be calculated subtracting the total urine collected from the total liquid consumed
Net Fluid Balance | 240 minutes after beverage consumption
  Net fluid balance will be calculated subtracting the total urine collected from the total liquid consumed
Urine Osmolality | 0 minutes before beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 0 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 60 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 120 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 180 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 240 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Sodium | 0 minutes before beverage consumption
  Urine Sodium will be measure in millimoles per liter.
Urine Sodium | 0 minutes after beverage consumption
  Urine Sodium will be measure in millimoles per liter.
Urine Sodium | 60 minutes after beverage consumption
  Urine Sodium will be measure in millimoles per liter.
Urine Sodium | 120 minutes after beverage consumption
  Urine Sodium will be measure in millimoles per liter.
Urine Sodium | 180 minutes after beverage consumption
  Urine Sodium will be measure in millimoles per liter.
Urine Sodium | 240 minutes after beverage consumption
  Urine Sodium will be measure in millimoles per liter.
Urine Potassium | 0 minutes before beverage consumption
  Urine Potassium will be measure in millimoles per liter.
Urine Potassium | 0 minutes after beverage consumption
  Urine Potassium will be measure in millimoles per liter.
Urine Potassium | 60 minutes after beverage consumption
  Urine Potassium will be measure in millimoles per liter.
Urine Potassium | 120 minutes after beverage consumption
  Urine Potassium will be measure in millimoles per liter.
Urine Potassium | 180 minutes after beverage consumption
  Urine Potassium will be measure in millimoles per liter.
Urine Potassium | 240 minutes after beverage consumption
  Urine Potassium will be measure in millimoles per liter.
Urine Specific Gravity | 150 minutes before beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 0 minutes before beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 0 minutes after beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 60 minutes after beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 120 minutes after beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 180 minutes after beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 240 minutes after beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Body Mass | 0 minutes before beverage consumption
  Body Mass in kilograms will be measured using a digital scale.
Body Mass | 240 minutes after beverage consumption
  Body Mass in kilograms will be measured using a digital scale.
Mood and Digestive Questionnaire | 0 minutes before beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 0 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 60 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 120 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 180 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 240 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Diastolic Blood Pressure | 0 minutes before beverage consumption
  Diastolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Diastolic Blood Pressure | 0 minutes after beverage consumption
  Diastolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Diastolic Blood Pressure | 60 minutes after beverage consumption
  Diastolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Diastolic Blood Pressure | 120 minutes after beverage consumption
  Diastolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Diastolic Blood Pressure | 180 minutes after beverage consumption
  Diastolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Diastolic Blood Pressure | 240 minutes after beverage consumption
  Diastolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Systolic Blood Pressure | 0 minutes before beverage consumption
  Systolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Systolic Blood Pressure | 0 minutes after beverage consumption
  Systolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Systolic Blood Pressure | 60 minutes after beverage consumption
  Systolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Systolic Blood Pressure | 120 minutes after beverage consumption
  Systolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Systolic Blood Pressure | 180 minutes after beverage consumption
  Systolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Systolic Blood Pressure | 240 minutes after beverage consumption
  Systolic Blood Pressure will be measured in millimeters mercury using an automated cuff.
Heart Rate | 0 minutes before beverage consumption
  Heart rate will be measured in beats per minute using an automated cuff.
Heart Rate | 0 minutes after beverage consumption
  Heart rate will be measured in beats per minute using an automated cuff.
Heart Rate | 60 minutes after beverage consumption
  Heart rate will be measured in beats per minute using an automated cuff.
Heart Rate | 120 minutes after beverage consumption
  Heart rate will be measured in beats per minute using an automated cuff.
Heart Rate | 180 minutes after beverage consumption
  Heart rate will be measured in beats per minute using an automated cuff.
Heart Rate | 240 minutes after beverage consumption
  Heart rate will be measured in beats per minute using an automated cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States